CLINICAL TRIAL: NCT01978808
Title: A Prospective Multi-center Randomized Study of the Difference in Diagnostic Yield Between EUS-FNA Needles With and Without a Side Port in Pancreatic Masses
Brief Title: Efficiency Study of the EUS-FNA Needles With and Without a Side Port in Pancreatic Masses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201307045RINC
Record Dates: First submitted 2013-10-16; First posted 2013-11-08 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatic Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
For diagnosis of pancreatic tumors, endoscopic ultrasound (EUS) and EUS-guided fine needle aspiration (EUS-FNA) are well established techniques in clinical practice. We hypothesize that a FNA needle with a side port could improve the diagnostic yield. The aim of this prospective randomized study is to determine whether there is a difference in diagnostic yield in patients with pancreatic masses for evaluation.

DETAILED DESCRIPTION:
For diagnosis of pancreatic tumors, endoscopic ultrasound (EUS) and EUS-guided fine needle aspiration (EUS-FNA) are well established techniques in clinical practice. In the case of EUS, an ultrasonic transducer located at the tip of the echoendoscope allows the endoscopist to visualize the wall of gastrointestinal tract as a series of definable layers corresponding to histology, and also enables detailed images of areas outside of the digestive tract. EUS has a significant clinical impact because it allows assessment of submucosal GI lesions, loco-regional staging of gastrointestinal malignancy, tissue diagnosis by EUS-FNA and staging of pancreaticobiliary lesions, non-small-cell lung carcinoma, and mediastinal disease. In prospective trials, EUS-FNA has been clearly established to be an important diagnostic tool with excellent safety profile.

Olympus has recently made commercially available a new 22 gauge FNA needle with a side port at the needle tip to facilitate the process of FNA and increase the diagnostic yield. There have been preliminary unpublished retrospective data that suggested the yield might be raised. However, there are no prospective multicenter randomized controlled studies to ascertain the validity of the assumption. The aim of this prospective randomized study is to determine whether there is a difference in diagnostic yield between EZ-Shot 2 (model: NA-220H-8022) and EZ-Shot 2 with side port (NA-230H-8022) in patients with pancreatic masses for evaluation. We hypothesize that a FNA needle with a side port could improve the diagnostic yield.

ELIGIBILITY:
Inclusion criteria:

1. all patients referred for EUS-FNA of pancreatic masses;
2. informed consent is obtained for performance of EUS-FNA.

Exclusion criteria:

1. presence of active gastrointestinal bleeding

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred for EUS-FNA of pancreatic masses
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
the overall diagnostic accuracy rate of both needles | assessment of diagnostic accuracy rate after 26 wks, then annually later

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Yao Cheng, Principal Investigator — Visiting staff
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan